CLINICAL TRIAL: NCT04764955
Title: Effect of Maternal Vitamin D3 Supplementation on Iron Status During Pregnancy and Early Infancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Bill and Melinda Gates Foundation (Other); King's College London (Other)
Responsible Party: Principal Investigator, Daniel Roth, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1000061108
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Pregnancy
Keywords: Maternal Nutrition; Vitamin D; Iron Status; Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A (Placebo) (Placebo Comparator): Prenatal Period 0 IU/week (17-24 weeks gestation - delivery) ; Postpartum Period 0 IU/week (delivery-6 months postpartum)
  Interventions: Dietary Supplement: Placebo
- Group B (4200:0 IU/week) (Experimental): Prenatal Period 4200 IU/week (17-24 weeks gestation - delivery) ; Postpartum Period 0 IU/week (delivery-6 months postpartum)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Vitamin D3 (cholecalciferol)
- 16800:0 IU/week (Experimental): Prenatal Period 16800 IU/week (17-24 weeks gestation - delivery) ; Postpartum Period 0 IU/week (delivery-6 months postpartum)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Vitamin D3 (cholecalciferol)
- 28000:0 IU/week (Experimental): Prenatal Period 28000 IU/week (17-24 weeks gestation - delivery) ; Postpartum Period 0 IU/week (delivery-6 months postpartum)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Vitamin D3 (cholecalciferol)
- 28000:28000 IU/week (Experimental): Prenatal Period 28000 IU/week (17-24 weeks gestation - delivery) ; Postpartum Period 28000 IU/week (delivery-6 months postpartum)
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)

INTERVENTIONS:
Dietary Supplement: Placebo — This product is identical in appearance, taste and texture to the experimental formulation but does not include any vitamin D3.
  Arms: 16800:0 IU/week; 28000:0 IU/week; Group A (Placebo); Group B (4200:0 IU/week)
Dietary Supplement: Vitamin D3 (cholecalciferol) — The intervention is an oral tablet containing vitamin D3 (cholecalciferol). Each weekly dose consists of a single tablet. Vitamin D3 content of the dose depends on the intervention group.
  Arms: 16800:0 IU/week; 28000:0 IU/week; 28000:28000 IU/week; Group B (4200:0 IU/week)

SUMMARY:
This is a secondary-use study based on previously-collected data and blood samples from a previously completed double-blind, dose-ranging trial of maternal prenatal and postpartum vitamin D supplementation in Dhaka, Bangladesh (NCT01924013). The aim of this sub-study is to examine the effect of vitamin D supplementation on iron status during pregnancy and early infancy.

DETAILED DESCRIPTION:
The risk of both low iron and vitamin D status have been recognized as public health concerns among pregnant women and young children, with high rates of deficiency in low-and middle-income countries. Through its involvement in regulation of the hepcidin-ferroportin axis, as well as its potential to increase the expression of the erythropoietin receptor, vitamin D has been suggested as a modulator of iron homeostasis. Vitamin D supplementation may therefore represent a candidate facilitator for the management of iron deficiency, yet few intervention trials have directly assessed the effect of vitamin D supplementation on biomarkers of iron status.

To examine the effect of vitamin D supplementation on iron status during pregnancy and early infancy, data and blood samples will be drawn from a completed double-blind, dose-ranging trial of maternal prenatal and postpartum vitamin D supplementation. Women at 17-24 weeks' gestation were randomized to 1 of 5 dose groups comprising a prenatal; postpartum regimen of placebo; placebo, 4200;0, 16800;0, 28000;0 or 28000;28000 IU vitamin D3/week until 26 weeks postpartum. Enrolment (n=1300) was completed in September 2015, and all infants were delivered by February 2016. The MDIG trial was primarily designed to determine the effect of maternal vitamin D on infant length at 12 months of age (with follow-up continuing until infants reached 24 months of age; completed in March 2018).

Analyses of serum ferritin and related iron biomarkers (serum iron, transferrin, soluble transferrin receptor, hepcidin), and inflammatory makers (e.g. CRP), will be conducted using previously collected stored blood samples. Linear regression models will be used to assess the effect of vitamin D supplementation on the biomarkers of interest among pregnant women and their infants at 6 months of age.

To examine the potential dose-response relation between prenatal vitamin D treatment dose (i.e., across all 4 assigned prenatal vitamin D doses by combining the 2 high-dose prenatal vitamin D treatment groups) and the biomarker of interest, linear regression models will be fitted using the assigned prenatal vitamin D treatment group as the categorical exposure variable and the specified biomarker as the (continuous) outcome variable. Data will be reported as mean differences (or mean % differences, if applicable) and 95% CIs.

To explore potential effects of prenatal only versus prenatal plus postpartum vitamin D supplementation on Hb and ferritin concentrations among infants at 6 months of age, a similar dose-response analysis will be conducted across all 5 treatment groups (i.e., disaggregation of the 2 high-dose prenatal vitamin D groups), for which the investigators will regress the biomarker (Hb as a continuous variable) on the vitamin D treatment group assigned during the prenatal and postpartum periods (as a categorical variable). Differences in each supplementation group will therefore be compared to the placebo group, and expressed as mean differences (or geometric means, or mean % differences, if applicable) and 95% CIs.

Given the influence of inflammation on serum ferritin concentrations, secondary analyses will include inflammatory markers (e.g. CRP) as covariates to test the role of inflammation in mediating the association between the vitamin D intervention and serum ferritin concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and above.
* Gestational age of 17 to 24 completed weeks estimated based on recalled last menstrual period (LMP) and/or ultrasound.
* Intends to permanently reside in the trial catchment area for at least 18 months
* MDIG trial participants with availability of at least one measurement of the biomarkers of interest (serum ferritin, circulating hepcidin, transferrin, soluble transferrin receptor, serum iron and/or whole-blood Hb).

Exclusion Criteria:

* History of medical conditions that may predispose the participant to vitamin D sensitivity, altered vitamin D metabolism and/or hypercalcemia, or history of renal calculi.
* High-risk pregnancy based on one or more of the following findings by point-of-care testing:
* - Severe anemia: hemoglobin <70 g/L assessed by Hemocue.
* - Moderate-severe proteinuria: ≥ 300 mg/dl (3+ or 4+) based on urine dipstick.
* - Hypertension: systolic blood pressure ≥140 mm Hg and/or diastolic blood pressure ≥90 mm Hg.
* - Multiple gestation, major congenital anomaly, or severe oligohydramnios based on maternal history and/or ultrasound.
* - Unwillingness to stop taking non-study vitamin D or calcium supplements or a multivitamin with calcium and/or vitamin D.
* - Currently prescribed vitamin D supplements as part of a physician's treatment plan for vitamin D deficiency.
* - Previous participation in the same study.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Maternal serum ferritin concentration at delivery | Delivery
  Maternal serum ferritin concentration at delivery

SECONDARY OUTCOMES:
Maternal transferrin saturation at delivery | Delivery
  Maternal transferrin saturation at delivery
Maternal soluble transferrin receptor at delivery | Delivery
  Maternal soluble transferrin receptor at delivery
Maternal circulating hepcidin at delivery | Delivery
  Maternal circulating hepcidin at delivery
Infant whole-blood Hb concentration | 6 months of age
  Infant whole-blood Hb concentration at 6 months of age
Infant ferritin concentration | 6 months of age
  Infant ferritin concentration at 6 months of age
Maternal total iron binding capacity at delivery | Delivery
  Maternal total iron binding capacity at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Roth, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- See also: Primary trial registration (MDIG) — https://www.clinicaltrials.gov/ct2/show/NCT01924013